CLINICAL TRIAL: NCT01891786
Title: A Randomised Control Trial (RCT) to Investigate the Effectiveness of a Selfmanagement Intervention and Personalised Genetic Risk Information to Reduce Risk of Coronary Heart Disease in Patients With Type 2 Diabetes.
Brief Title: Coronary Heart Disease Risk in Type 2 Diabetes
Acronym: CORDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Stanton Newman, Professor, City, University of London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12/EE/0437; RRMR11-001 (Other Grant/Funding Number: The Bupa Foundation)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Heart Disease; Type 2 Diabetes
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): The participant's General practitioner (GP) practice and/or practice nurse will provide care as normal for their patient.
- Group Self-Management Intervention (SMI) (Active Comparator): Participants will be asked to attend a total of 4 SMI sessions delivered on a weekly basis.
  Interventions: Behavioral: Self-Management Intervention
- SMI + Risk Results (Active Comparator): The participant will provide a saliva sample for analysis. They will attend an appointment with their nurse to receive personalised results on their combined genetic and lifestyle risk for developing CHD in the next 10 years. They will then be asked to attend the 4 week SMI programme.
  Interventions: Behavioral: Self-Management Intervention; Behavioral: Risk Result

INTERVENTIONS:
Behavioral: Self-Management Intervention — The SMI will incorporate a discussion to introduce self-management and why it is important, and about problems associated with reducing CHD risk and managing type 2 diabetes. Specific topics addressed will include health behaviours to reduce CHD risk and manage diabetes including diet and exercise, as well as behaviours specific to managing diabetes, including medication adherence and self-care behaviours (e.g. footcare). Sessions are patient-directed and employ a shared decision-making approach, such that participants work with one another and the practice nurse facilitator to identify specific problems that they wish to address, and to identify solutions and approaches to managing their diabetes and CHD risk
  Arms: Group Self-Management Intervention (SMI); SMI + Risk Results
Behavioral: Risk Result — Participants will receive in-person personalised feedback about their combined genetic and lifestyle 10 year risk for developing CHD.
  Arms: SMI + Risk Results

SUMMARY:
The primary objective of the CORDIA study is to use an effective evidence-based self-management intervention (SMI) for type 2 diabetes, with and without a novel test to give a personalised genetic and lifestyle risk of coronary heart disease, to examine their capacity to reduce the risk of coronary heart disease (CHD) and improve diabetes management in primary care patients with type 2 diabetes. The effect of these interventions on clinical, behavioural and psychological outcomes will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 25-70 years diagnosed with type 2 diabetes
* White, Afro-Caribbean or Asian-Indian ethnicity
* Most previous or baseline HbA1c ≥6.5% or 48 mmol/mol
* Fluency in written and spoken English

Exclusion Criteria:

* Diagnosis of ischemic heart disease, stroke, Transient Ischaemic Attack (TIA) or peripheral vascular disease
* Serious or enduring mental health problems that would prevent the patient from completing the study
* Currently receiving treatment for a life-threatening condition (e.g., cancer) or in the terminal stages of a condition
* Adults who cannot consent for themselves

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Coronary heart disease 10 year risk | 12 months
  Coronary heart disease 10 year risk as assessed using the United Kingdon Prospective Diabetes Study (UKPDS) Risk Calculator

SECONDARY OUTCOMES:
Psycho-social impact of the intervention | 12 months
  Psycho-social impact of the intervention conditions will be assessed using questionnaires designed to measure risk perception, self-efficacy, and motivation. Feelings of anxiety and depression will also be assessed.
Health behaviour impact of the intervention | 12 months
  The impact of the intervention conditions on health behaviours including diet, exercise and smoking behaviour will be assessed in addition to a range of diabetes self-care behaviours such as foot care and blood glucose self-monitoring.
Impact of receiving genetic results | 6 months
  The impact of receiving genetic test results using a modified version of the Multidimensional Impact of Cancer Risk Assessment (MICRA) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Stanton P Newman, PhD, Principal Investigator — City, University of London
Locations (10):
- United Kingdom (10):
  - Addison House Surgery, Harlow, Essex
  - Church Street Surgery, Ware, Essex
  - Dolphin House Surgery, Ware, Essex
  - Wallace House Surgery, Hertford, Hertfordshire
  - Cambridgeshire Community Services NHS Trust, Cambridgeshire
  - Chesterfield Drive Surgery, Ipswich
  - Martlesham health Surgery, Ipswich
  - Dr Taylor and Partners, Woodbridge Suffolk
  - The Peninsula Practice, Woodbridge Suffolk
  - Wickham Market Medical Centre, Woodbridge Suffolk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beaney KE, Ward CE, Bappa DA, McGale N, Davies AK, Hirani SP, Li K, Howard P, Vance DR, Crockard MA, Lamont JV, Newman S, Humphries SE. A 19-SNP coronary heart disease gene score profile in subjects with type 2 diabetes: the coronary heart disease risk in type 2 diabetes (CoRDia study) study baseline characteristics. Cardiovasc Diabetol. 2016 Oct 3;15(1):141. doi: 10.1186/s12933-016-0457-7. PMID 27716211
- [Derived] Davies AK, McGale N, Humphries SE, Hirani SP, Beaney KE, Bappa DA, McCabe JG, Newman SP. Effectiveness of a self-management intervention with personalised genetic and lifestyle-related risk information on coronary heart disease and diabetes-related risk in type 2 diabetes (CoRDia): study protocol for a randomised controlled trial. Trials. 2015 Dec 2;16:547. doi: 10.1186/s13063-015-1073-7. PMID 26631181